CLINICAL TRIAL: NCT06288633
Title: Cardioneuroablation for Bradyarrhythmia (Sinus Node and Atrioventricular Node Dysfunction): a Sham-controlled Randomised Multicentre Trial
Brief Title: Cardioneuroablation for Bradyarrhythmia
Acronym: CARDIOBOOST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Collaborators: Meshalkin National Medical Research Center, Ministry of Health of Russian Federation (Other Government); The Federal Centre of Cardiovascular Surgery, Russia (Other); Clinical City Hospital named after I.V. Davydovsky of Moscow Department of Healthcare (Network); City Clinical Hospital No.52 of Moscow Healthcare Department (Other); National Medical Research Center for Therapy and Preventive Medicine (Other Government); Medical Centre Hospital of the President's Affairs Administration, Republic of Kazakhstan (Other Government); Tomsk National Research Medical Center of the Russian Academy of Sciences (Other); Vishnevsky Center of Surgery (Other); National Medical Research Center for Cardiology, Ministry of Health of Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FNWMRC
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Bradycardia; Syncope; Sick Sinus Syndrome
Keywords: bradycardia; cardioneuroablation; sinus node dysfunction; atrioventricular node dysfunction
MeSH Terms: conditions — Bradycardia; Syncope; Sick Sinus Syndrome | interventions — Electrophysiologic Techniques, Cardiac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardioneuroablation (Active Comparator): Radiofrequency catheter transmyocardial ablation of the ganglion plexuses (GP) of the atria - cardioneuroablation. The procedure is performed under local anesthesia using intracardiac catheters. Radiofrequency applications will be applied to the endocardial surface of the left and/or right atria in places of typical localization of the densest GPs network in order to destroy nerve fibers and ganglia: in patients with sinus bradycardia - in the left and right atria (5 places with the highest concentration of ganglia); in patients with impaired atrioventricular conduction - in the right atrium and in the left atrium (1 place in the right atrium - at the ostium of the coronary sinus; 2 places in the left atrium - opposite the ostium of the coronary sinus and opposite the Marshall ligament/vein).
  Interventions: Procedure: Ganglionated plexi ablation
- Sham group (Sham Comparator): In the control (sham) group, endocardial electrophysiological study will be performed, but patients will not know which procedure they performed (they are "blinded" in relation to the distribution group). The monitoring will be performed according to the same protocol as in the cardioneuroablation group. In case of recurrence of symptomatic bradycardia and/or (with) syncopal condition without traumatization of the patient in the control group, a transition to the cardioneuroablation group (cross-over) will be proposed. In case of disagreement, a pacemaker is implanted.
  Interventions: Diagnostic Test: Electrophysiological study

INTERVENTIONS:
Procedure: Ganglionated plexi ablation — Through access in the femoral vein, a mapping or ablation-mapping catheter is inserted into the right atrium, and a three-dimensional reconstruction of the right atrium is performed using an electroanatomic mapping system. The inferior and superior vena cava, the coronary sinus are indicated.
  Then a transeptal puncture is performed using a transeptal introducer and a needle for transeptal puncture under fluoroscopic control. A three-dimensional reconstruction of the left atrium is performed using an electroanatomic mapping system.
  During or immediately after the creation of three-dimensional maps of both atria, areas of the typical concentration of ganglion plexuses (GP) are ablated using radiofrequency applications (30-50 Watts, 10-40 s each point). Ablated points are annotated on the three-dimensional map. GPs ablation zones are about 0.5 x 1.0 cm in size.
  Arms: Cardioneuroablation
Diagnostic Test: Electrophysiological study — Through access in the femoral vein, a diagnostic catheter is inserted in the area of the coronary sinus under fluoroscopic control. The effective refractory period (ERP) of the atria will be measured according to the method adopted in clinical practice, namely: using a ten-pole diagnostic electrode installed in the coronary sinus, a series of eight electrical pulses with the same amplitude and frequency is applied to the atrial myocardium. Then the ninth pulse is applied with a gradual decrease in the time interval until the absence of an atrial myocardium response to the pulse is registered. The cycle of an additional, ninth pulse, in which the atrial myocardium did not respond to an electrical impulse, is considered an atrial ERP.
  Arms: Sham group

SUMMARY:
This is a multicenter prospective randomized blind controlled trial with a sham procedure group of the efficacy and safety of cardioneuroablation as a method of treating symptomatic bradycardia without a permanent pacemaker implantation

DETAILED DESCRIPTION:
Catheter ablation is a common treatment for cardiac arrhythmias. Some patients with AF ablation or AVNRT experience acceleration of sinus rhythm, the most likely cause of which is modification of autonomic tone caused by inadvertent damage to intramural autonomic ganglia and fibers. Intentional damage to these plexuses has become known as cardioneuroablation (CNA) and is currently used in patients with tachycardia-bradycardia syndrome, vegetatively caused sinus node dysfunction and atrioventricular conduction disorders, vasovagal syncopal conditions developing in a cardioinhibitory type.

It is suggested that in some patients CNA may become an alternative to permanent pacemaker for the treatment of symptomatic bradyarrhythmias.

This is a multicentre randomised clinical study evaluating the efficacy of cardioneuroablation for severe bradycardia due to sinus node dysfunction and/or atrioventricular nide dysfunction versus a sham procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Any of the following variants of bradyarrhythmia in patients aged 18-65 years:

   (1.1.) Symptomatic sinus bradycardia or bradycardia due to atrioventricular blockade, including transient.

   (1.2.) Severe asymptomatic sinus bradycardia with a rhythm frequency of <30 beats/min.

   (1.3.) Transient atrioventricular block of II-III degree or permanent block of II degree.

   (1.4.) Repeated fainting or pre-fainting states with a proven association with bradycardia (without injury).

   (1.5.) Rhythm pauses >6 seconds.

   In combination with the following two criteria:
2. Positive reaction to physical activity and/or atropine test:

   (2.1.) Increase in sinus rhythm frequency ≥25% or >90 beats/min. (2.2.) The transition of atrioventricular blockade of the II-III degree to the 1st degree or complete normalization of atrioventricular conduction at the sinus rhythm.
3. Sinus rhythm at the time of switching on

Exclusion Criteria:

1. Anamnesis of injury during syncopation due to bradycardia, except in the case when the patient refused to implant an electrocardiostimulator for his own reasons in writing;
2. Constant intake of antiarrhythmic drugs (for PVC, AF, etc.);
3. The presence of an implanted pacemaker, a heart contractility modulation device, a cardioverter defibrillator;
4. Drug-induced sinus bradycardia and/or atrioventricular block;
5. Bradycardia due to electrolyte imbalance (e.g. hyperkalemia);
6. Bradycardia due to hypothyroidism or other reversible conditions;
7. No reaction to the administration of atropine (up to a maximum dose of 0.2 mg / kg);
8. Proven association of bradyarrhythmia with episodes of apnea/hypopnea in obstructive sleep apnea syndrome;
9. Clinically significant coronary artery disease;
10. Postinfarction cardiosclerosis;
11. Hemodynamically significant congenital heart defects, including operated ones;
12. Stroke or transient ischemic attack <3 months;
13. Open heart surgery in the anamnesis;
14. Catheter interventions on coronary arteries or for cardiac arrhythmias <3 days;
15. Conditions after percutaneous coronary angioplasty <3 months;
16. Anamnesis of stable ventricular tachycardia on the background of bradycardia;
17. Pregnancy or breastfeeding period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Implantation of a permanent cardiac pacemaker | 12 months post procedure
  Once there is a recurrence of documented symptomatic bradycardia, a permanent pacemaker implantation is considered

SECONDARY OUTCOMES:
Complications of cardioneuroablation | 30 days post procedure
  Cardiac tamponade, pericardial effusion >10 mm, esophageal damage, stroke or transient ischemic event, severe groin hematoma (hemoglobin level drop >20%), atriovenous fistula in the groin
Presence of symptomatic or asymptomatic rhythm pauses >6 seconds | 12 months post procedure
  As detected by ECG monitoring
The presence of symptomatic or asymptomatic sinus bradycardia with an average heart rate <40 beats/min in the daytime | 12 months post procedure
  As detected by ECG monitoring
Transient or permanent atrioventricular block | 12 months post procedure
  As detected by ECG monitoring
Orthostatic hypotension and/or bradycardia during passive orthostasis test | 12 months post procedure
  Tilt-testing
Sinus tachycardia after cardioneuroablation | 30 days post procedure
  As detected by ECG monitoring, defined as daytime mean heart rate >100 bpm
Implantation of a pacemaker by 24 months after randomization | 24 months post procedure
  Once there is a recurrence of documented symptomatic bradycardia, a permanent pacemaker implantation is considered

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Mikhaylov, Prof., Principal Investigator — Almazov National Medical Research Centre
Locations (1):
- Almazov National Medical Research Centre, Saint Petersburg, Russia